CLINICAL TRIAL: NCT07204093
Title: Transdermally Applied Estradiol Delivery In Ultra-Safe Medications Valuable In Treatment Against Endometriosis
Brief Title: Ultra-Safe Hormonal Strategy: Transdermal Estradiol Added to Progestins for Endometriosis
Acronym: TAEDIUMVITAE
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 0021423-U; TAEDIUMVITAE (Other: Comitato Etico Territoriale Lombardia 3)
Record Dates: First submitted 2025-09-08; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-07

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — drospirenone; dienogest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with endometriosis undergoing medical management: This cohort will include women of reproductive age with a confirmed diagnosis of endometriosis, either by laparoscopy/histology or by validated imaging techniques (e.g., transvaginal ultrasound, MRI).
  Interventions: Drug: Drospirenone 4 mg orally; Drug: Dienogest 2 mg orally

INTERVENTIONS:
Drug: Drospirenone 4 mg orally — Daily oral administration of Drospirenone 4 mg + Transdermal estradiol; continuous administration for at least 6 months.
  Other Names: Slinda
Drug: Dienogest 2 mg orally — Daily oral administration of Dienogest 2 mg + Transdermal estradiol; continuous administration for at least 6 months.
  Other Names: Visanne; Dienogest; Zafrilla

SUMMARY:
Endometriosis is a chronic, estrogen-dependent disease affecting women of reproductive age, associated with pelvic pain, infertility, and reduced quality of life. Progestins are the standard first-line therapy, but long-term treatment requires well-tolerated regimens that balance efficacy with patient satisfaction.

This study will compare two combinations of progestins with natural transdermal estradiol-dienogest versus drospirenone-to evaluate which regimen provides greater patient satisfaction after 6 months of therapy.

DETAILED DESCRIPTION:
Endometriosis is a chronic, estrogen-dependent disorder characterized by the presence of endometrial tissue outside the uterine cavity. This ectopic tissue induces chronic inflammation, fibrosis, and adhesions, often resulting in pelvic pain, dysmenorrhea, dyspareunia, infertility, and impaired quality of life. The condition affects an estimated 6-10% of women of reproductive age, with peak prevalence between 25 and 35 years, making it one of the most common gynecological diseases with significant social and economic impact.

Available treatments for endometriosis are symptomatic rather than curative. Medical management is considered the cornerstone of therapy, especially in women who are not seeking immediate pregnancy. Current guidelines recommend progestins as first-line treatment due to their proven efficacy in suppressing endometriosis-associated pain and their favorable safety and tolerability profile. However, because therapy is usually long-term until menopause and continuous, optimal regimens must combine efficacy with good tolerability and sustained patient satisfaction.

Dienogest is an established fourth-generation progestin widely used in endometriosis management, with well-documented efficacy and safety. Drospirenone, another fourth-generation progestin, combines progestogenic, anti-androgenic, and anti-mineralocorticoid activities. Although marketed primarily as a contraceptive, drospirenone has shown promising results in controlling endometriosis symptoms and improving patient-reported outcomes.

Progestin-only regimens may lead to hypoestrogenic adverse effects, including vaginal dryness, mood disturbances, reduced libido, irregular bleeding, and bone loss. For this reason, the addition of natural estradiol is considered advantageous, as it may prevent atrophic changes, support bone metabolism, and improve overall quality of life. Transdermal estradiol, in particular, avoids hepatic first-pass metabolism, does not induce prothrombotic liver factors, and is associated with a lower risk of thromboembolic events compared with ethinyl estradiol.

This observational study is designed to directly compare two therapeutic strategies for women with endometriosis: Dienogest + transdermal estradiol or Drospirenone + transdermal estradiol.

The primary endpoint is patient satisfaction after 6 months of treatment, reflecting the central importance of patient-centered outcomes in a chronic disease that impacts multiple aspects of daily life. Secondary endpoints include sexual function, psychological well-being, and health-related quality of life, assessed with validated questionnaires.

By comparing two modern progestin-based regimens combined with natural estradiol, this study aims to generate evidence that will help clinicians tailor hormonal therapy to improve not only symptom control but also the long-term well-being and quality of life of women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* women who have been on combination therapy for at least 6 months with progestin and transdermal natural oestrogen (Dienogest + transdermal oestradiol or Drospirenone + transdermal oestradiol);
* women who have performed follow-up at least 6 months after the start of treatment and for whom data on the primary endpoint of the study (treatment satisfaction) are available.

Exclusion Criteria:

* absence of surgical diagnosis or imaging indicative of endometriosis or adenomyosis;
* women who have taken GnRH analogue therapy within 6 months prior to treatment with dienogest + transdermal oestradiol vs. drospirenone + transdermal oestradiol
* women who have taken only progestogen therapy without transdermal oestradiol or with contraindications to oestrogen use;
* women who received surgical indications during the treatment period, including obstructive uropathy or symptomatic bowel stricture; evidence of complex ovarian cysts or ovarian endometriomas with a diameter greater than 5 cm on transvaginal ultrasound.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with endometriosis referred to the endometriosis outpatient clinic of the Gynaecology SC of the Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico in Milan between October 2024 and September 2025 will be included in the study. The diagnosis of endometriosis is made on the basis of the combination of symptomatology + gynaecological examination, transvaginal/transrectal ultrasound or previous surgical visualisation of the disease.
Sampling Method: Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Patients' statisfaction | This outcome will be evaluated after at least 6 months of treatment
  Therapy satisfaction will be assessed by means of a 5-level Likert scale (very satisfied; satisfied; neither satisfied nor dissatisfied; dissatisfied; very dissatisfied). Women expressing the judgement 'very satisfied' and 'satisfied' will be considered to be globally satisfied, similarly to reported in the study on which the calculation of the sample size is based. The outcome will be dichotomised (very satisfied + satisfied versus neither satisfied nor dissatisfied + dissatisfied + very dissatisfied).
  The level of statisfaction in the two groups will be compared as the proportion of satisfied women in each treatment group, reported as frequencies and percentages and analyzed accordingly.

SECONDARY OUTCOMES:
Therapeutic efficacy - symptoms control (NRS) | This outcome will be evaluated after at least 6 months of treatment
  Symptoms control, measured by Numeric Rating Scale (NRS), 11-point (0 = no pain; 10 = worst imaginable pain) for the following symptoms: dysmenorrhea, deep dyspareunia, superficial dyspareunia, non-menstrual pelvic pain, pain during defecation, pain during urination.
Therapeutic efficacy - symptoms control (use of analgesics) | This outcome will be evaluated after at least 6 months of treatment
  Symptoms control, measured by use of analgesic therapy for pain symptoms, as reported during clinical evaluation (0 = no, 1 = yes).
Therapeutic efficacy - ovulation suppression | This outcome will be evaluated after at least 6 months of treatment
  Confirmation of ovulation suppression, the therapeutic goal in endometriosis management, through serum measurement of 17β-estradiol, progesterone, and follicle-stimulating hormone (FSH), according to clinical practice.
Therapeutic efficacy - amenorrhea achievement and bleeding pattern | This outcome will be evaluated after at least 6 months of treatment
  Bleeding pattern during treatment, with number achieving amenorrhea (therapeutic goal in endometriosis medical management). Unexpected uterine bleeding will be recorded as: spotting, menstrual-like bleeding, or heavy bleeding. The cumulative number of bleeding days and the number of treatment interruptions lasting one week (tailored cycling) to manage irregular bleeding will be collected.
Global Impression of Change | This outcome will be evaluated after at least 6 months of treatment
  Patients' Global Impression of Change (PGIC) Scale, single-item, 7-point Likert scale (very much improved; much improved; minimally improved; no change; minimally worse; worse; very much worse).
Sexual function | This outcome will be evaluated after at least 6 months of treatment
  Measured by the Female Sexual Function Index (FSFI), 19-item questionnaire with 5-point Likert scale. The final score will be interpreted as continuous (lower scores indicating worse sexual function)
Mood changes | This outcome will be evaluated after at least 6 months of treatment
  Measured by the Hospital Anxiety and Depression Scale (HADS), 14-item, 4-point Likert scale. The total score will be interpreted as continuous (lower scores indicating better psychological status).
Health-related quality of life (HRQoL) | This outcome will be evaluated after at least 6 months of treatment
  Calculated using the 12-Item Short Form Health Survey (SF-12) questionnaire, with Physical Component Summary (PCS-12) and Mental Component Summary (MCS-12). The total score will be interpreted as continuous (lower scores indicating worse health status).
Acceptance of transdermal therapy | This outcome will be evaluated after at least 6 months of treatment
  Measured by:
  * 11-point numeric scale (0 = no discomfort; 10 = worst imaginable discomfort).
  * 5-level categorical scale (1 = no discomfort; 5 = intolerable discomfort).
Adverse events | This outcome will be evaluated after at least 6 months of treatment
  Assessed globally through a single-item question on side effects reported during treatment (as previously used in the sample size reference study). Reported side effects will be collected, and, if present, their impact on quality of life will be evaluated using a 10-point numeric scale (1 = minimal impact; 10 = maximum impact).
Treatment adherence | This outcome will be evaluated after at least 6 months of treatment
  Measured by the Morisky Medication-Taking Adherence Scale (MMAS-4), single-item, with scores ranging from 0 = excellent adherence to 4 = poor adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecology Unit, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided